CLINICAL TRIAL: NCT01631773
Title: A Comparison of microRNA Samples in Patients With Nasal Polyps and Aspirin Exacerbated Respiratory Disease and Those With Nasal Polyps Only
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Dennis Ledford, Principal Investigator, University of South Florida
Other Study IDs: Nasal Polyp Study & Aspirin
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Aspirin-exacerbated Respiratory Disease; Nasal Polyp
Keywords: Aspirin-exacerbated respiratory disease; Nasal polyp
MeSH Terms: conditions — Nasal Polyps | interventions — MicroRNAs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal epithelial tissue will be collected from the inferior nasal turbinates of ten subjects with nasal polyps and AERD disease and from the inferior turbinates of ten subjects with nasal polyps but without AERD. A rhinoprobe™ will be used to collect this epithelial tissue. These samples will be analyzed by miRNA assay to determine if there is a difference in mircroRNA expression between the two subject groups.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- subjects w/ Nasal polyps & AERD disease: subjects with nasal polyps and Aspirin-exacerbated respiratory disease (AERD) disease
  Interventions: Genetic: microRNA
- subjects w/ nasal polyps without AERD: subjects with nasal polyps but without Aspirin-exacerbated respiratory disease (AERD)
  Interventions: Genetic: microRNA

INTERVENTIONS:
Genetic: microRNA — Biological samples will be taken from subjects w/ Nasal polyps & AERD disease and subjects w/ nasal polyps without AERD. MicroRNA will be analyzed to compare genetic similarities and differences between the two study groups.

SUMMARY:
We hypothesize that the miRNA expression in subjects with nasal polyps and Aspirin-exacerbated respiratory disease (AERD) differs from the miRNA expressed in subjects with nasal polyps but without Aspirin-exacerbated respiratory disease (AERD).

DETAILED DESCRIPTION:
Nasal epithelial tissue will be collected from the inferior nasal turbinates of ten subjects with nasal polyps and AERD disease and from the inferior turbinates of ten subjects with nasal polyps but without AERD. A rhinoprobe™ will be used to collect this epithelial tissue. These samples will be analyzed by miRNA assay to determine if there is a difference in mircroRNA expression between the two subject groups.

ELIGIBILITY:
Inclusion Criteria:

* Ages eligible for study: 18 to 70 years
* Genders eligible for study: male and female
* Signed and dated written informed consent is obtained prior to study
* Subjects have a physician diagnosis of nasal polyps without AERD or physician diagnosis of nasal polyps with AERD. The diagnosis of aspirin sensitive asthma must be present for a minimum of three months. If the medical history is indeterminate either an aspirin challenge will be required to confirm or rule out the diagnosis. An aspirin challenge is a protocol that can safely be performed as an out patient procedure with close supervision.

Exclusion Criteria:

* Pregnant and/or lactating females.
* Current tobacco use.
* Severe psychiatric illness.
* Current illicit substance use or dependence and/or abuse of alcohol.
* Primary or secondary immunodeficiency.
* Any clinically significant uncontrolled medical condition that would put the patient at risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be a prospective study design with a target sample size of 20. The objective of conducting it as a prospective study is to confirm that the sampling procedures and analysis methodology work as expected before attempting a larger study. We propose to have 10 study participants with nasal polyps but without AERD and 10 study participants with nasal polyps and AERD. If the results of this study are promising, larger studies with sufficient power for statistical analysis will be considered.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Positibe Group: 2 fold or greater will be identified as differntially expressed MiRNA. | No time frame noted
  5 total groups
Negative Group: MiRNAs are absent from both groups | No time frame noted
  5 total groups

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Ledford, MD, Principal Investigator — Division of Allergy and Immunology, Department of Internal Medicine, University of South Florida College of Medicine
Locations (1):
- USF Division of Allergy and Clinical Immunology Clinical Research Unit, Tampa, Florida, United States